CLINICAL TRIAL: NCT00004042
Title: A Phase I Dose-Escalation Study of BIBH-1 in Patients With Advanced or Metastatic Fibroblast Activation Protein-Positive Cancer
Brief Title: Monoclonal Antibody F19 in Treating Patients With Advanced or Metastatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: BOEH-1152.1; MSKCC-98068; CDR0000066903 (Registry Identifier: PDQ (Physician Data Query)); LUDWIG-LUD98-002; NCI-H99-0025
Record Dates: First submitted 1999-12-10; First posted 2004-08-20 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2009-12

CONDITIONS: Colorectal Cancer
Keywords: stage III colon cancer; stage IV colon cancer; stage III rectal cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms

INTERVENTIONS:
Biological: monoclonal antibody F19
Radiation: iodine I 131 monoclonal antibody F19

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Phase I trial to study the effectiveness of monoclonal antibody F19 in treating patients who have advanced or metastatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Identify the toxicity associated with increasing doses of monoclonal antibody F19 (BIBH-1) administered weekly by intravenous infusion in patients with unresectable, advanced or metastatic fibroblast activation protein-positive colorectal cancer. II. Determine the dose limiting toxicity and maximum tolerated dose of this drug in these patients. III. Measure induction titers of human anti-human antibody to BIBH-1 and correlate immunologic-related clinical effects. IV. Determine the pharmacokinetics, biodistribution, and imaging characteristics of increasing intravenous doses of the drug. V. Document tumor responses in this patient population.

OUTLINE: This is a dose escalation, open label, multicenter study. Patients receive monoclonal antibody F19 (BIBH-1) IV over 60 minutes weekly for 12 weeks. The first, fifth, and ninth treatments are combined with iodine I 131. Patients with stable or responding disease may continue treatment for up to 12 months. The dose of BIBH-1 is escalated in cohorts of 3-6 patients until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose limiting toxicity. Patients are followed at 1 month.

PROJECTED ACCRUAL: A maximum of 24 patients will be accrued for this study within 8 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed unresectable, advanced and/or metastatic disease: Colorectal cancer Measurable or evaluable disease Epidemiologically proven fibroblast activation protein positive Failed or refused conventional treatment, and unlikely to derive significant benefit from conventional treatments No active CNS metastases No new or progressive lesions on CT scan, more than 3 months since treatment (i.e., surgery or radiotherapy) for brain metastases, and/or not receiving mitomycin Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 18 and over Menopausal status: Not specified Performance status: Karnofsky 70-100% Life expectancy: At least 4 months Hematopoietic: Absolute granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: ALT/AST no greater than 3 times upper limit of normal Bilirubin less than 2 mg/dL Renal: Creatinine no greater than 2.0 mg/dL Other: Not pregnant or nursing Fertile patients must use effective contraception No other serious illness No active infections requiring antibiotics No bleeding disorders No other diseases that may potentially interfere with obtaining accurate study results

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior immunotherapy No prior murine, chimeric or humanized antibody and/or antibody fragment Chemotherapy: See Disease Characteristics At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas and mitomycin) Endocrine therapy: No concurrent systemic corticosteroids (except for acute management of allergic-type events) No concurrent immunosuppressive agents Radiotherapy: See Disease Characteristics Surgery: See Disease Characteristics Recovered from surgery Other: At least 4 weeks since other prior investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 1998-11; Primary Completion 2001-07 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sydney Welt, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (2):
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Memorial Sloan-Kettering Cancer Center, New York, New York
- Ludwig Institute for Cancer Research-Sydney Branch, Sydney, New South Wales, Australia